CLINICAL TRIAL: NCT02823314
Title: Effectiveness of Medical Taping Concept Applied in the T7-T8 Dermatome in Nausea and Vomiting After Chemotherapy in Cancer Patients
Brief Title: Effectiveness of Medical Taping Concept in Cancer Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Hospital Universitario San Juan de Alicante (Other)
Responsible Party: Principal Investigator, María Isabel Tomás-Rodríguez, PT, Doctor, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16/308
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Cancer-related Problem/Condition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): One piece of a special hypoallergenic adhesive tape, called Cure Tape®, they will have a size of 12-20 cm and will be attached in the front and back torso area on the T7- T8 dermatomes.
  Interventions: Device: Cure Tape™ covering T 7 and T 8 dermatomes
- Placebo group (Placebo Comparator): Two piece of a special hypoallergenic adhesive tape, called Cure Tape®, have a size of 2.5 cm x 2 cm and they will have to be placed near the greater trochanter area.
  Interventions: Device: Cure Tape™ away from dermatomes T 7 and T 8

INTERVENTIONS:
Device: Cure Tape™ covering T 7 and T 8 dermatomes — The intervention group will have to apply two strips of special hypoallergenic tape called Cure Tape™ that will have a size of 20 x 5 cm and they will have to be placed on the T7-T8 dermatome area.
  Other Names: Kinesio Taping
  Arms: Intervention group
Device: Cure Tape™ away from dermatomes T 7 and T 8 — The control group will have to apply two strips of special hypoallergenic tape called Cure Tape™ that will have a size of 5 x 4 cm and they will have to be placed near the greater trochanter area.
  Other Names: Kinesio Taping
  Arms: Placebo group

SUMMARY:
Nausea and vomiting are two of the side effects associated with the most common antineoplastic chemotherapy treatments. The Medical Taping Concept (MTC) is an economical technique, easy to apply. This is a technique that may help reduce nausea and vomiting after application of chemotherapy in cancer patient.

DETAILED DESCRIPTION:
Nausea and vomiting are two of the side effects associated with the most common antineoplastic chemotherapy treatments. There are some studies that support the use of physical measures such as TENS or acupuncture to lessen these effects.

The Medical Taping Concept (MTC) is an economical technique, easy to apply and few side effects. In some manuals on this technique the possibility that it may act to reduce nausea and vomiting described. Sim But after a comprehensive literature search have not found jobs to support these assumptions. With this work, the research team will attempt to obtain evidence on the effects of its application in the areas of influence of the dermatome T7 and T8. For this, two adhesive tapes of this type of bandage is placed on the front and back on a group of patients after receiving chemotherapy session and compared with a control group that will apply this technique outside the dermatome indicated . Both groups will receive antiemetics according to the service routine. If the hypothesis were positive it could extend the application of this simple technique to cancer patients from other centers in order to help reduce nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Neoadjuvant and adjuvant breast cancer
* To have been diagnosed with a severe comorbid disorder
* To have received at least the first cycle of emetogenic chemotherapy

Exclusion Criteria:

* Not suffer nausea or vomiting episodes in the previous cycle of chemotherapy,
* To Shower inability to report nausea and / or vomiting.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-10 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Difference between Number of times you have vomited during the first 24 hours after the first chemotherapy session and after the second chemotherapy session | 24 hours after the first chemotherapy session and 24 hours after the second chemotherapy session
  1, 2, 3, 4, 5, .........
Difference between nausea after the first chemotherapy session and after the second chemotherapy session | 24 hours after the first chemotherapy session and 24 hours after the second chemotherapy session
  Nausea (Yes / No)
Difference between Intensity of nausea in the experience of the participant after the first chemotherapy session and after the second chemotherapy sessionintervention and pre-intervention | 24 hours after the first chemotherapy session and 24 hours after the second chemotherapy session
  numerical scale from 0 to 10 (0 = No / 10 = maximum)

SECONDARY OUTCOMES:
Difference between Quality of life post-intervention and pre-intervention | 24 hours after chemotherapy and 4 days after chemotherapy
  EQ-5D™ is a standardised instrument for use as a measure of health outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de San Juan, Sant Joan DÁlacant, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Spanish law: 15/1999 Data Protection

REFERENCES:
- [Background] Chao LF, Zhang AL, Liu HE, Cheng MH, Lam HB, Lo SK. The efficacy of acupoint stimulation for the management of therapy-related adverse events in patients with breast cancer: a systematic review. Breast Cancer Res Treat. 2009 Nov;118(2):255-67. doi: 10.1007/s10549-009-0533-8. PMID 19760035
- [Background] Ezzo J, Richardson MA, Vickers A, Allen C, Dibble S, Issell BF, Lao L, Pearl M, Ramirez G, Roscoe JA, Shen J, Shivnan JC, Streitberger K, Treish I, Zhang G, Manheimer E. WITHDRAWN: Acupuncture-point stimulation for chemotherapy-induced nausea or vomiting. Cochrane Database Syst Rev. 2014 Nov 21;(11):CD002285. doi: 10.1002/14651858.CD002285.pub3. No abstract available. PMID 25412832
- [Background] Gardani G, Cerrone R, Biella C, Galbiati G, Proserpio E, Casiraghi M, Arnoffi J, Meregalli M, Trabattoni P, Dapretto E, Giani L, Messina G, Lissoni P. A progress study of 100 cancer patients treated by acupressure for chemotherapy-induced vomiting after failure with the pharmacological approach. Minerva Med. 2007 Dec;98(6):665-8. PMID 18299681
- [Background] Huertas-Fernandez MJ, Martinez-Bautista MJ, Sanchez-Martinez I, Zarzuela-Ramirez M, Baena-Canada JM. [Analysis of the effectiveness of an antiemetic protocol used in an oncology division]. Farm Hosp. 2010 May-Jun;34(3):125-38. doi: 10.1016/j.farma.2009.11.001. Spanish. PMID 20206564
- [Background] Abdel-Kadar M. Percutaneous Electrical Neurostimulation (PENS) of Dermatome T6 with an Ambulatory Self-applied Patch vs PENS of Dermatome T6 with Conventional Procedure: Effect on Appetite and Weight Loss in Moderately Obese Patients. Obes Surg. 2016 Dec;26(12):2899-2905. doi: 10.1007/s11695-016-2214-0. PMID 27289457
- [Background] Tomas-Rodriguez MI, Palazon-Bru A, Martinez-St John DRJ, Toledo-Marhuenda JV, Asensio-Garcia MDR, Gil-Guillen VF. Effectiveness of medical taping concept in primary dysmenorrhoea: a two-armed randomized trial. Sci Rep. 2015 Nov 13;5:16671. doi: 10.1038/srep16671. PMID 26564807
- See also: Newsletters kinesiology-tape — http://www.kineweb.es/articulos-kinesiology-tape-vendaje-neuromuscular.html
- See also: Newsletters Medical Taping concept — http://www.aneid.com/about-us/background